CLINICAL TRIAL: NCT05026073
Title: Application of Vibrational Biospectroscopy as a Novel Diagnostic Tool in Endometrial Cancer
Brief Title: Vibrational Spectroscopy for Endometrial Cancer Diagnosis
Acronym: SPEED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19ON033
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Endometrial Cancer; Endometrial Hyperplasia
Keywords: endometrial cancer; uterine neoplasm; cancer of the endometrium; Spectroscopy; Raman spectroscopy; Fourier Transform Infrared spectroscopy; endometrial hyperplasia
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia; Uterine Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be retained for the duration of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 Endometrial Cancer:: Women with histological diagnosis of cancer of the endometrium (any type) undergoing hysterectomy
  Interventions: Behavioral: Information about clinical risk factors for endometrial cancer and endometrial hyperplasia; Procedure: Blood and endometrial tissue sampling; Procedure: Lymph node sampling
- Group 2 Endometrial Hyperplasia:: Women with histological diagnosis of endometrial hyperplasia (with or without atypia) undergoing hysterectomy
  Interventions: Behavioral: Information about clinical risk factors for endometrial cancer and endometrial hyperplasia; Procedure: Blood and endometrial tissue sampling
- Group 3 Controls:: Healthy women undergoing hysterectomy for a benign reason
  Interventions: Behavioral: Information about clinical risk factors for endometrial cancer and endometrial hyperplasia; Procedure: Blood and endometrial tissue sampling

INTERVENTIONS:
Behavioral: Information about clinical risk factors for endometrial cancer and endometrial hyperplasia — age, race, parity, body mass index, last menstrual period, menstrual cycle type, hypertension, type II diabetes, anovulation, polycystic ovary syndrome, indication for hysterectomy and smoking history. Other epidemiologic risk factors including tamoxifen exposure, history of breast cancer, current hormone therapy use, anticoagulant use, oral contraception use, family history of endometrial, breast or colon cancer.
Procedure: Blood and endometrial tissue sampling — * All women will undergo planned hysterectomy.
  * Venous blood sample will be collected prior to surgery.
  * Endometrial sampling via Pipelle device will be performed immediately prior to hysterectomy
  * Endometrial biopsy from the hysterectomy specimen will be obtained under direct vision
  The plasma and serum obtained from the blood samples will be analysed with ATR-FTIR and Raman spectroscopes. Spectra from both wet and dry specimens will be recorded.
  All tissue samples retrieved will be placed in Phosphate Buffered Solution for transfer to the histopathology laboratory. Spectra will be collected from the fresh samples with ATR-FTIR and Raman spectroscopes. Spectral analyses will subsequently be repeated on dry samples post fixation and processing.
  All tissue samples will undergo haematoxylin and eosin staining after spectral analysis for standard histopathological confirmation.
Procedure: Lymph node sampling — Lymph nodes will be excised if recommended as part of the standard treatment for endometrial cancer.
  Each node will be cut in half or in quarters, depending on size, to expose the core. Wet and dry spectral analysis will be performed, followed by staining for histopathological confirmation.
  Groups: Group 1 Endometrial Cancer:

SUMMARY:
The purpose of this study is to investigate the ability of vibrational spectroscopic techniques, Raman spectroscopy and Attenuated Total Reflection - Fourier Transform Infrared spectroscopy (ATR-FTIR), to accurately differentiate endometrial tissue, lymph nodes and blood samples with womb cancer or endometrial hyperplasia from healthy controls.

DETAILED DESCRIPTION:
Womb cancer is the sixth most common cancer in women, with rising incidence worldwide. Current diagnostic strategies are time consuming, invasive and have limited accuracy, furthermore there is no population-wide screening. Treatment depends on patients' health, type of disease and spread at the time of diagnosis. Most women will be offered surgery, however the role of lymph node dissection in early stage disease remains controversial.

There is therefore a need for an objective, accurate test, able to detect pre-cancer and cancer early and able to identify metastatic node involvement, so that lymph node excision is performed only when necessary.

Attenuated Total Reflection - Fourier Transform Infrared (ATR-FTIR) spectroscopy and Raman spectroscopy are non-invasive, objective techniques that use the interaction of light within tissues to gain detailed information about the chemical composition of biological samples. These methods have shown tremendous potential for improving diagnosis and treatment of cancer.

This study aims to use Vibrational Spectroscopy to examine blood plasma and serum, endometrial biopsies via Pipelle device and pelvic/para-aortic lymph nodes for the presence of endometrial pre-cancer and cancer changes. The analyses will be performed on fresh (wet) as well as dried samples.

The ultimate goal is to develop a point-of-care test and an intra-operative tool for endometrial cancer screening and diagnosis. Such a test could speed up endometrial cancer diagnosis, reduce treatment delays and individualise patients care.

ELIGIBILITY:
Inclusion Criteria:

1. Endometrial cancer group:

   * Established histopathological diagnosis of cancer of the endometrium (any stage and subtype)
   * Patients must be eligible for primary staging surgery (any route, e.g. laparoscopy and laparotomy)
2. Endometrial hyperplasia group:

   * Established histopathological diagnosis of endometrial hyperplasia (with or without atypia)
   * Treatment with hysterectomy deemed necessary
3. Control group

   * Healthy with benign disease, non-malignancy
   * Undergoing hysterectomy (any route, e.g. laparoscopy and laparotomy)

Exclusion Criteria:

* Patient's refusal / inability to consent
* Synchronous gynaecological cancer (ovary, cervix, fallopian tubes)
* Previous pelvic radiotherapy
* Previous hysterectomy
* Undiagnosed vaginal bleeding
* Previous endometrial ablation

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women undergoing hysterectomy with a histological diagnosis of primary cancer of the endometrium (irrespective of subtype), or endometrial hyperplasia (with or without atypia) and women undergoing hysterectomy for a benign indication.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-01-19 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Vibrational Spectroscopy diagnostic accuracy | Baseline
  The primary outcome of the study will be to evaluate the correct classification of cases of endometrial cancer, endometrial hyperplasia and controls by Raman and ATR-FTIR spectral analysis, compared to histopathology as the standard of reference. The outcome will be measured with sensitivity, specificity, positive/negative predictive values and likelihood ratios.
  The diagnostic accuracy will be documented for pipelle samples, endometrial samples from hysterectomy specimens, pelvic/para-aortic lymph nodes, blood serum and plasma.

SECONDARY OUTCOMES:
Discriminating wavenumbers | Baseline
  Identification of the most important wavenumbers that distinguish between normal, hyperplasia and cancer
Sub-analysis of endometrial cancer and hyperplasia sub-types | Baseline
  sub-analysis of segregation percentages for pre-cancerous changes (non-atypical / atypical hyperplasia) and cancer subtypes
Test reliability | Baseline
  Calculation of inter- and intra- user classification variability
Multivariate analysis of patient and tumour characteristics | Baseline
  Multivariate analysis of variance will be calculated to account for factors potentially affecting test performance (histological subtype, menopausal status, age, co-morbidities, hormonal treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Ketankumar Gajjar, MD, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, England, United Kingdom